CLINICAL TRIAL: NCT03550092
Title: Application of Graph Theory to Both Resting-state and Task-based fMRI Data to Uncover Brain-behavior Relationships Related to Therapy Outcomes in Aphasia
Brief Title: Analysis of Brain Activity to Uncover Brain-behavior Relationships Related to Therapy Outcomes in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Chaleece Sandberg, Assistant Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DC016708-01A1 (NIH)
Record Dates: First submitted 2018-05-11; First posted 2018-06-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Aphasia
Keywords: aphasia; treatment; therapy; anomia; fMRI; neuroimaging; semantics
MeSH Terms: conditions — Aphasia; Anomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aphasia (Experimental): Abstract Semantic Association Network Training (AbSANT) Each session will be 2 hours long and will occur twice each week for a total of 20 sessions.
  Interventions: Behavioral: Abstract Semantic Association Network Training (AbSANT)

INTERVENTIONS:
Behavioral: Abstract Semantic Association Network Training (AbSANT) — In each session, the participant will be asked to categorize words, choose/discuss semantic features for each word that accurately describe the word, and generate as many words as possible within a category.
  Other Names: Semantic word-finding therapy; Semantic Feature Analysis/Verification

SUMMARY:
Aphasia is a loss of language due to stroke or other brain injury. Word-finding in conversation is a universal and persistent difficulty in aphasia. While several techniques exist to improve word-finding in aphasia, it is unclear how the brain changes in response to behavioral therapy. In this study, persons with aphasia will receive behavioral therapy aimed at helping them to be more successful at finding words. Twenty therapy sessions will be provided in a 10-week period. Each therapy session will last about 2 hours and will include a variety of language tasks. Prior to beginning word-finding therapy, each participant will receive two fMRI scans, spaced 10 weeks apart. After finishing therapy, each participant will receive two additional fMRI scans, spaced 10 weeks apart. For a portion of the MRI scan, participants will complete language tasks. The purpose of these fMRI scans is to measure brain changes that may occur due to successful behavioral therapy. The hypotheses are as follows: First, that the behavioral therapy will improve word-finding as it has been shown to do in the past. Second, that the brain will change in a couple of different ways. It is expected that the network of regions that support word-finding will be more connected and work together more efficiently after therapy. It is also expected that the networks of regions that support other aspects of cognitive function, such as attention and executive function, will also be more connected and work together more efficiently.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of aphasia
2. Sustained stroke more than 6 months prior to consent
3. Right-handed
4. Native speakers of English
5. Completed at least a high school education
6. Normal or corrected-to-normal vision and hearing
7. Provide written informed consent
8. Participants will be medically stable and at least wheelchair ambulatory at the time of participation with uncompromised use of the left hand

Exclusion Criteria:

1. History of degenerative neurological disorders (e.g., Alzheimer's disease), acquired neurological disorders other than aphasia from stroke (e.g., traumatic brain injury), developmental neurological disorders (e.g., autism), or psychiatric disorders
2. An active medical condition that could compromise participation (e.g., cancer undergoing acute treatment)
3. Not safe to enter the bore of the magnet (e.g., pacemaker)
4. Taking medications that are known to exert significant effects on cognitive processes
5. Pregnancy or possibility of pregnancy
6. Do not meet the above inclusionary criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Therapy Effect Size: Change in word generation performance from pre- to post-treatment measured using a version of Cohen's d | At baseline and at approximately 10 weeks (i.e., the end of therapy)
  The mean of the baseline scores is subtracted from the mean of the post-treatment scores, and then divided by the standard deviation (SD) of the baseline scores. 6.5-8 is considered a small effect size, 8-9.5 is medium, and above 9.5 is large.
Change in fMRI activation patters from pre- to post-treatment | At baseline and at approximately 10 weeks (i.e., the end of therapy)
  Blood-oxygen-level-dependent MRI signal measured during task and rest and subjected to statistical tests of significant change from pre- to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chaleece W Sandberg, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Hershey Medical Campus, Hershey, Pennsylvania, United States